CLINICAL TRIAL: NCT00684385
Title: An International Expanded Access Clinical Programme With ZD1839 (IRESSA) for Patients With Advanced Non-small Cell Lung Cancer(NSCLC) and Patients With Recurrent or Metastatic or Both Recurrent and Metastatic Squamous Cell Carcinoma of the Head and Neck (H&NC)
Brief Title: An Expanded Access Programme With Iressa for Patients With Non-Small-Cell Lung Cancer and Cancer of the Head and Neck
Status: Approved for marketing | Type: Expanded Access
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: 1839IL/0052; D7914C00052
Record Dates: First submitted 2008-05-21; First posted 2008-05-26 (Estimated); Last update posted 2019-03-14 (Actual); Status verified 2019-02

CONDITIONS: Non Small Cell Lung Cancer; Cancer of the Head and Neck
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Head and Neck Neoplasms | interventions — Gefitinib

STUDY DESIGN:
Expanded Access Types: Individual

INTERVENTIONS:
Drug: ZD1839 — 250mg administered daily for patients with NSCLC and500mg daily for patients with H&NC. Treatment dispensed to patients on Day 1 and every 12 weeks thereafter until the patient withdraws. Patients with NSCLC will take one tablet at each dose administration; patients with squamous cell H&NC will take two tablets at each dose administration.
  Other Names: Iressa

SUMMARY:
The purpose of this study is to provide ZD1839 for those patients with locally advanced and/or metastatic non-operable non-small cell lung cancer (stage III or IV) or recurrent and/or metastatic squamous cell head and neck cancer who receive the therapy on an expanded access basis due to their inability to meet eligibility criteria for on-going recruiting trials, inability to participate in other clinical trials (e.g., poor performance status, lack of geographic proximity), or because other medical interventions are not considered appropriate or acceptable.

ELIGIBILITY:
Inclusion Criteria:

* Have received at least one course of standard systemic chemotherapy or radiation therapy
* Are ineligible for chemotherapy or radiotherapy
* Are ineligible or not candidates for enrollment in available ZD1839 trials for NSCLC or squamous cell H&NC
* Are, in the investigators opinion, not medically suitable for chemotherapy.

Exclusion Criteria:

* Current eligibility (i.e., meeting the inclusion and exclusion criteria except signed informed consent) for any ZD1839 protocol available to the patient, or previous enrollment in a blinded ZD1839 protocol
* Patients from a blinded protocol may be considered for acceptance, with AstraZeneca's permission, only after trial completion and unblinding of all patients.
* Patients eligible for or previously enrolled in an open-label or unblinded ZD1839 clinical trial may be considered for acceptance with AstraZeneca's permission
* Incomplete healing from prior oncologic or other major surgery

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Yuri Rukazenkov, Study Director — AstraZeneca
Locations (27):
- Germany (20):
  - Research Site, Berlin
  - Research Site, Essen
  - Research Site, Frankfurt
  - Research Site, Freiburg im Breisgau
  - Research Site, Göttingen
  - Research Site, Großhansdorf
  - Research Site, Halle
  - Research Site, Heidelberg
  - Research Site, Kiel
  - Research Site, Laatzen
  - Research Site, Lemgo
  - Research Site, Löwenstein
  - Research Site, Mainz
  - Research Site, München
  - Research Site, Nuremberg
  - Research Site, Oldenburg
  - Research Site, Stralsund
  - Research Site, Stuttgart
  - Research Site, Trier
  - Research Site, Wiesbaden
- Hungary (3):
  - Research Site, Budapest
  - Research Site, Kecskemét
  - Research Site, Törökbálint
- Poland (3):
  - Research Site, Gdansk
  - Research Site, Warsaw
  - Research Site, Zabrze
- Research Site, Newcastle upon Tyne, United Kingdom